CLINICAL TRIAL: NCT03250754
Title: Treatment of Headache Disorders With Acupuncture: Observational Study (HDACU)
Brief Title: Treatment of Headache Disorders With Acupuncture: Observational Study: OBSERVATIONAL STUDY (HDACU)
Acronym: HDACU
Status: Completed | Type: Observational
Sponsor: Hospital Son Llatzer (Other)
Responsible Party: Principal Investigator, Javier Mata, Chief of Section of Anesthesiology and Reanimation Department, Hospital Son Llatzer
Other Study IDs: HDACU-001
Record Dates: First submitted 2017-08-11; First posted 2017-08-16 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Chronic Headache Disorder
Keywords: Acupuncture; Migraine; Tension-type headache
MeSH Terms: conditions — Migraine Disorders; Tension-Type Headache | interventions — Electroacupuncture

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pharmacological treatment group: Treatment decision making is based on physician's choice and patient preferences. Patients were referred to the Pain Service Unit. Patients continued with a prophylactic treatment alone
- Electroacupuncture group: Treatment decision making is based on physician's choice and patient preferences. Patients were referred to the Pain Service Unit. Patients continued with a new prophylactic treatment and additionally, received 12 sessions of acupuncture. The treatments, which included electro-stimulation.
  Interventions: Device: Electroacupuncture

INTERVENTIONS:
Device: Electroacupuncture — Needles on the extremities were stimulated by electro-stimulation device applied by a biphasic pulse generator apparatus at a frequency of pulses alternated between 2 Hz and 100 Hz and the maximum tolerable intensity.
  Groups: Electroacupuncture group

SUMMARY:
Headache disorders (HDs), which are characterized by recurrent headache, constitute a public-health problem of enormous proportions, with an impact on both the individual sufferer and society. The stated goals of long-term headache treatment are to reduce the frequency, severity, and disability associated with acute attacks; decrease the reliance on poorly tolerated, ineffective, or unwanted acute pharmacotherapies; and avoid acute headache medication escalation. There is risk for adverse events, leading some patients to refuse prophylactic therapy. Acupuncture is widely used for the treatment of headaches and it may be applied as a single modality as well as part of a more complex treatment program. The objective of this study will be to investigate whether acupuncture in routine clinical practice ((Real World Data) is more effective than treatment of acute migraine attacks or routine care only in reducing headache frequency.

DETAILED DESCRIPTION:
A Cochrane systematic review published in 2016 concluded that acupuncture was at least as effective as, or possibly more effective than, preventive drug treatment for migraine prophylaxis with fewer side effects compared with conventional treatments . Cochrane reviews of tension-type headache conclude that acupuncture could be a valuable non-pharmacological tool in patients with frequent, episodic, and chronic tension-type headache.

An observational, cross-sectional study, according to the STROBE guide, was conducted. The study was carried out in the Pain Service Unit of the Son Llàtzer University Hospital of Palma de Mallorca, Spain.

Between January 2010 and December 2015, data from patients with chronic refractory headache, which did not respond to conventional treatment for at least 6 months, referred to the Pain Service Unit were examined to ascertain their eligibility.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of headache (> 12 months) and at least two headaches per month (Physicians classified patients according to the criteria of the International Headache Society to differentiate between patients with, tension-type headache, trigeminal autonomic cephalgias (cluster headache and Horton's headache), trigeminal neuralgia, occipital neuralgia, cervicogenic headache and post-surgery headache).
* Age ≥ 18 years.

Exclusion Criteria:

* Headache caused by somatic diseases such as hypertension, meningioma or meningoencephalitis
* Onset of headache less than 1-year before.
* acupuncture treatment less than 1-year before

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with headache disorder, which did not respond to conventional treatment for at least 6 months, referred to the Pain Service Unit were examined to ascertain their eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 482 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Number of days with headache per month | At the end of the third month of treatment
  Because the improvements observed were essentially proportional to the headache at study entry, we also calculated the percent reduction of headache days for each patient. Treatment responders were also calculated: a patient with a reduction of ≥ 50% was considered to be a treatment responder.

SECONDARY OUTCOMES:
Visual analogue scale (VAS) for pain | at baseline, 1 month and 3-months
  a continuous scale comprised of a horizontal line, anchored by "no pain" (score of 0) and "worst imaginable pain" (score of 100 [100-mm scale]). (VAS pain intensity score)
The change of headache days after 1 month | at baseline, 1 month and 3-months
  Number of headache days per month
Assessment of satisfaction with treatment | at baseline, 1 month and 3-months
  ranging from 10 (extremely Satisfied) to 0 (extremely dissatisfied)
Sleep quality assessment | at baseline, 1 month and 3-months
  ranging from 10 (good quality) to 0 (poor quality)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Mata, MD, Principal Investigator — Son Llatzer University Hospital
Locations (1):
- Son Llàtzer University Hospital, Palma, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: Undecided
No later than 3 years after the study will have ended a completely deidentified data set will deliver to an appropriate data archive for sharing purposes

REFERENCES:
- [Background] Headache Classification Subcommittee of the International Headache Society. The International Classification of Headache Disorders: 2nd edition. Cephalalgia. 2004;24 Suppl 1:9-160. doi: 10.1111/j.1468-2982.2003.00824.x. No abstract available. PMID 14979299
- [Background] Garcia-Escriva A, Asensio-Asensio M, Lopez-Hernandez N, Gonzalez-Aznar OJ, Oliver-Navarrete C, Alvarez-Sauco M, Pampliega-Perez A. [Health care activity in a headache-specific clinic]. Rev Neurol. 2004 Sep 1-15;39(5):401-5. Spanish. PMID 15378449
- [Background] Linde K, Allais G, Brinkhaus B, Fei Y, Mehring M, Vertosick EA, Vickers A, White AR. Acupuncture for the prevention of episodic migraine. Cochrane Database Syst Rev. 2016 Jun 28;2016(6):CD001218. doi: 10.1002/14651858.CD001218.pub3. PMID 27351677
- [Background] Linde K, Allais G, Brinkhaus B, Fei Y, Mehring M, Shin BC, Vickers A, White AR. Acupuncture for the prevention of tension-type headache. Cochrane Database Syst Rev. 2016 Apr 19;4(4):CD007587. doi: 10.1002/14651858.CD007587.pub2. PMID 27092807
- [Background] Vickers AJ, Cronin AM, Maschino AC, Lewith G, MacPherson H, Foster NE, Sherman KJ, Witt CM, Linde K; Acupuncture Trialists' Collaboration. Acupuncture for chronic pain: individual patient data meta-analysis. Arch Intern Med. 2012 Oct 22;172(19):1444-53. doi: 10.1001/archinternmed.2012.3654. PMID 22965186
- [Background] Wang LP, Zhang XZ, Guo J, Liu HL, Zhang Y, Liu CZ, Yi JH, Wang LP, Zhao JP, Li SS. Efficacy of acupuncture for acute migraine attack: a multicenter single blinded, randomized controlled trial. Pain Med. 2012 May;13(5):623-30. doi: 10.1111/j.1526-4637.2012.01376.x. Epub 2012 Apr 26. PMID 22536889
- [Background] Li Y, Liang F, Yang X, Tian X, Yan J, Sun G, Chang X, Tang Y, Ma T, Zhou L, Lan L, Yao W, Zou R. Acupuncture for treating acute attacks of migraine: a randomized controlled trial. Headache. 2009 Jun;49(6):805-16. doi: 10.1111/j.1526-4610.2009.01424.x. Epub 2009 Apr 27. PMID 19438740
- [Background] Yang CP, Chang MH, Liu PE, Li TC, Hsieh CL, Hwang KL, Chang HH. Acupuncture versus topiramate in chronic migraine prophylaxis: a randomized clinical trial. Cephalalgia. 2011 Nov;31(15):1510-21. doi: 10.1177/0333102411420585. Epub 2011 Oct 21. PMID 22019576
- [Background] Coeytaux RR, Kaufman JS, Kaptchuk TJ, Chen W, Miller WC, Callahan LF, Mann JD. A randomized, controlled trial of acupuncture for chronic daily headache. Headache. 2005 Oct;45(9):1113-23. doi: 10.1111/j.1526-4610.2005.00235.x. PMID 16178942
- [Background] Wonderling D, Vickers AJ, Grieve R, McCarney R. Cost effectiveness analysis of a randomised trial of acupuncture for chronic headache in primary care. BMJ. 2004 Mar 27;328(7442):747. doi: 10.1136/bmj.38033.896505.EB. Epub 2004 Mar 15. PMID 15023830
- [Background] Witt CM, Reinhold T, Jena S, Brinkhaus B, Willich SN. Cost-effectiveness of acupuncture treatment in patients with headache. Cephalalgia. 2008 Apr;28(4):334-45. doi: 10.1111/j.1468-2982.2007.01504.x. PMID 18315686
- [Background] Vandenbroucke JP. When are observational studies as credible as randomised trials? Lancet. 2004 May 22;363(9422):1728-31. doi: 10.1016/S0140-6736(04)16261-2. No abstract available. PMID 15158638
- [Background] Concato J, Shah N, Horwitz RI. Randomized, controlled trials, observational studies, and the hierarchy of research designs. N Engl J Med. 2000 Jun 22;342(25):1887-92. doi: 10.1056/NEJM200006223422507. PMID 10861325
- [Background] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) Statement: guidelines for reporting observational studies. Int J Surg. 2014 Dec;12(12):1495-9. doi: 10.1016/j.ijsu.2014.07.013. Epub 2014 Jul 18. PMID 25046131